CLINICAL TRIAL: NCT00327366
Title: Effect of Bright Light on Sex Hormones and Ovulation in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Russian Academy of Medical Sciences (Other)
Responsible Party: Outside In
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: M-s3
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Last update posted 2009-10-19 (Estimated); Status verified 2009-10

CONDITIONS: Anovulation
Keywords: Menstrual Cycle; Light Therapy; Sex Hormones; Ovulation
MeSH Terms: conditions — Anovulation | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Light therapy

SUMMARY:
The study investigated whether bright artificial light may influence menstrual cycle and ovulation conclusively, and what underlying hormonal changes for this effect are.

DETAILED DESCRIPTION:
Several studies have shown a shortening of the menstrual cycle following light therapy in women with abnormally long menstrual cycles or with winter depression, which suggests that bright light may influence sex hormones and ovulation. The study was designed to investigate this possibility. Twenty-two women with slightly lengthened menstrual cycles and without clinically evident endocrine abnormalities completed a study lasting for two menstrual cycles separated by an off-protocol episode of at least 1 menstrual cycle. Bright light therapy was administered for a week at home during one experimental cycle, and dim light during another cycle (placebo-controlled, crossover, counter-balanced order). Daytime blood sampling and ultrasound scan were performed before and after a week of light therapy, on the ~7th and 14th days after menstruation onset. Ultrasound examination was repeated further to document ovulation. Serum was assayed for thyroid-stimulating hormone, prolactin, luteinizing hormone, follicle-stimulating hormone, and estradiol. The preliminary results were reported at the SLTBR meeting in June, 2005.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-40 years
* Mean menstrual cycle 28-38 days
* Good general health
* Generally normal sleep-wake regimen
* Motivated for free participation

Exclusion Criteria:

* Low cooperation
* Medications known to interfere with hormone release
* Clinically evident endocrine abnormalities including the signs of
* Hyperandrogenism
* Travel over several time zones during two months prior the study

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2003-09; Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin V. Danilenko, MD, Principal Investigator — Institute of Internal Medicine SB RAMS